CLINICAL TRIAL: NCT05320822
Title: A Pragmatic Rehabilitation Intervention to Supplement Progressive Return to Activity Following Mild Traumatic Brain Injury in Service Members (SMs): The Active Rehab Study
Brief Title: A Pragmatic Rehabilitation Intervention: The Active Rehab Study
Acronym: ARM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-2904; CDMRP-PT190088 (Other Grant/Funding Number: USAMRAA)
Record Dates: First submitted 2022-01-27; First posted 2022-04-11 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Concussion, Brain
Keywords: Concussion, Rehabilitation
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progressive Return to Activity (Group 1) (Active Comparator): The current practice, Progressive Return to Activity (PRA) based on Traumatic Brain Injury Center of Excellence (TBICoE) protocols, provides a framework for activity progression based on participant symptom reports and recovery. PRA TBICoE includes a graded approach for clinicians to return participants to pre-injury activities based on the severity of the participant symptoms with and without physical exertion.
  Interventions: Other: Progressive Return to Activity (Group 1)
- Active Rehab (Group 2) (Experimental): Active Rehab includes an adaptive paradigm based on personal characteristics, symptom presentation, and duty requirements that integrate with current progressive return to activity (PRA TBICoE) guidelines. Activity progressions consider the initial presentation and changes in participant status during treatment, with the goal of safely accelerating recovery. Severity and presence of symptoms will guide progression as reported by the participant.
  The intervention consists of 5 phases designed to facilitate an active approach to concussion rehabilitation. Phases are symptom stabilization, impairment reduction, activity integration, recovery acceleration, and military duty specific application. Participants complete phase specific activities under direction of a clinical professional, and progress upon meeting specific requirements.
  Interventions: Other: Active Rehab (Group 2)

INTERVENTIONS:
Other: Active Rehab (Group 2) — The Active Rehab protocol builds off of initial chief complaints and duty profile and addresses symptom control followed by a progressive and prescribed integration of activities to full return to duty that should be integrated with the current PRA TBICoE protocols. The specific activity areas in the intervention include low-intensity aerobic exercise that does not exacerbate symptoms, cognition, balance, visual/vestibular, and comfort/ general well-being.
  Participants can be progressed daily according to symptom limitations. At least 3-4 sessions each week are recommended based on a trial of sport-related mTBI and other interventions of this type concerning mTBI/concussion. During each phase, low level aerobic exercise that does not significantly exacerbate symptoms, such as nature walks, will be recommended. The additional activity types that may be chosen include cognitive, balance, visual/vestibular, and comfort/general well-being.
  Arms: Active Rehab (Group 2)
Other: Progressive Return to Activity (Group 1) — Participant will be asked to use symptoms to guide activity from the time of the injury until participant is asymptomatic. Once asymptomatic, participant will begin the PRA TBICoE clinical recommendation. During this time clinicians will document activities in each stage in addition to initial symptom checklist, stage of PRA CoE progression, activity parameters, percentage of rest during the session, participants rating of perceived exertion, and final symptom checklist, session satisfaction rating, and session feedback.
  Arms: Progressive Return to Activity (Group 1)

SUMMARY:
The strategic objective of this research line is to examine improving short- and long-term outcomes for soldiers following mild traumatic brain injury (mTBI). The technical objectives are to: 1) conduct a Phase 1 quasi-experimental pragmatic trial testing the potential benefit of provider directed active rehabilitation therapies ("Active Rehab") in accelerating return of injured soldiers back to active duty and improving cognitive and functional limitations following mTBI, and 2) operationalize and disseminate a clinical active rehabilitation algorithm for use in military settings. The central hypothesis is that an active rehabilitation algorithm in the context of the progressive return to activity will improve clinical and functional outcomes, including time to return to duty.

The Active Rehab intervention expands on progressive return to activity guidelines by providing activities that can be completed and progressed during Stage 1 of the progressive return to activity protocol, when the participant is at least 24 hours postinjury. Active Rehab includes an adaptive paradigm based on personal characteristics, symptom presentation, and duty requirements that integrate with current progressive return to activity guidelines. Activity progressions consider the initial presentation and changes in participant status during treatment, with the goal of safely accelerating recovery. Severity and presence of symptoms will guide progression: worse, same or better as reported by the participant.

DETAILED DESCRIPTION:
The study population will be soldiers stationed at Fort Bragg, North Carolina. Allocation to arm will be determined by time (preintervention/current practice (Group 1) vs. intervention/Active Rehab (Group 2)). The study will enroll and follow mild traumatic brain injuries in the study population, presenting to study targeted providers within 2 weeks following mild traumatic brain injury/concussion, over two 9 month periods (n=65 in each period for a total n=130 completing the protocol). Post-injury patient outcomes include military performance, physiological, clinical and psychological health outcomes. Study assessment timepoints include initial post-injury intake, 2-weeks post enrollment (as possible), asymptomatic, and clearance to return to duty. In the first 9-month period (Study Phase 1), the study will evaluate current progressive return to activity practices and patient outcomes following mild traumatic brain injury.

In the second 9-month period (Study Phase 2), soldier participants will complete the Active Rehab protocol. Active Rehab activities will be progressed based on participants' reported symptoms and duty profiles. The intervention will be delivered through provider and study staff education to participants. Outcomes will be compared between the two study phases (current practice vs. Active Rehab). Following data acquisition, investigators will utilize Machine Learning techniques to develop an adaptive clinical Active Rehab protocol for military settings (Study Phase 3). The algorithm will use serial measures of military performance, physiological function, clinical recovery, and psychological health status obtained at acutely and sequentially throughout treatment to direct best options for an individual's Active Rehab protocol progression.

ELIGIBILITY:
Inclusion Criteria:

* Current active duty military personnel stationed at Fort Bragg, North Carolina.
* Report to clinic/provider at Fort Bragg and available for recruitment within 2 weeks of mTBI injury date as indicated in medical record.
* Initial provider diagnosis of mTBI/concussion within 2 weeks of injury, confirmed via medical record.

Exclusion Criteria:

* Third mTBI/concussion in the past 12 months as indicated by the medical record and/or participant self-report.
* Symptoms clear at rest and exertion within 48 hours as indicated in medical record and or during study enrollment process.
* Moderate-Severe TBI, or TBI not meeting the criteria for mTBI as indicated by provider diagnosis.
* Polytrauma or other injuries preventing completion of initial study assessments in the 2-week window as indicated in initial screening/medical record.

TBI, per the funding opportunity announcement is defined as: "being caused by (1) a direct blow or impact to the head, (2) a penetrating head injury, or (3) an exposure to external forces such as blast waves that disrupt the function of the brain." For the proposed study, only those meeting the VA/Department of Defense severity criteria of mild (normal structural imaging, loss of consciousness 0-30 minutes, alteration of consciousness or mental state up to 24 hours, posttraumatic amnesia up to 24 hours, and Glasgow Coma Scale of 13-15) will be targeted.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Average days to full return to duty clearance | 1 to approximately 360 days
  Average number of days from injury to clearance to full return to duty (date return to duty as reported by participant when returned to duty with no limitations or restrictions minus date of injury)

SECONDARY OUTCOMES:
Average days to asymptomatic | 1 to approximately 240 days
  Average number of days from injury to asymptomatic, determined as when no neurobehavioral symptom inventory (NSI) symptom is greater than 1.
Heart Rate Variability (HRV) | up to approximately 346 days after intervention initiation
  Heart rate variability (HRV) will be assessed during seated (parasympathetic dominant) and standing (sympathetic dominant) conditions. The conditions will be assessed over three, five minute intervals. Twice when the participant is seated, and once while the participant is standing. Assessment of these conditions allows for assessment of response to a change in state. Assessed at: Initial visit (Baseline); determination of asymptomatic state (up to approximately 226 days after intervention initiation); clearance to full return to duty after intervention completion (up to approximately 346 days after intervention initiation).
Cognitive Status using the Military Acute Concussion Evaluation 2 (MACE 2) | up to approximately 346 days after intervention initiation
  The MACE 2 will be used to assess cognitive status after acute injury. The MACE 2 has demonstrated validity, reliability, and sensitivity to concussion. The MACE 2 is a multimodal tool that assists in the assessment and diagnosis of concussion. It contains sections on orientation, immediate memory, concentration, and delayed memory. The sum scores from all sections are used to calculate a total score. Total score ranges from 0-30. Assessed at: Initial visit (Baseline); 2 weeks after intervention initiation, determination of asymptomatic state (up to approximately 226 days after intervention initiation); clearance to full return to duty after intervention completion (up to approximately 346 days after intervention initiation).
Near point convergence (NPC) | up to approximately 346 days after intervention initiation
  Near-point convergence is a commonly used oculomotor exam that defines the amplitude of convergence or the closest point in space where the participant can hold fusion, and therefore, see one target. Participants complete 3 trials assessing near-point convergence, distance in centimeters, and the average of the three trials is recorded. Assessed at: Initial visit (Baseline); 2 weeks after intervention initiation, determination of asymptomatic state (up to approximately 226 days after intervention initiation); clearance to full return to duty after intervention completion (up to approximately 346 days after intervention initiation).
Coordination using the Balance Error Scoring System (BESS) Total Score | up to approximately 346 days after intervention initiation
  The Balance Error Scoring System (BESS) is a commonly used measure of static balance and postural stability. A combination of three stances (narrow double leg stance, single leg stance, and tandem stance) and two footing surfaces (firm surface/floor or medium density foam) are used for the test. Each stance is held, with hands on hips and eyes closed, for 20 seconds. Points are given for specific behaviors ("errors"), including opening eyes, lifting hands off hips, or stepping, stumbling or falling. Total score ranges from 0-60. Assessed at: Initial visit (Baseline); 2 weeks after intervention initiation, determination of asymptomatic state (up to approximately 226 days after intervention initiation); clearance to full return to duty after intervention completion (up to approximately 346 days after intervention initiation).
Neurobehavioral Symptom Inventory total score and individual symptom scores | up to approximately 346 days after intervention initiation
  The Neurobehavioral Symptom Inventory (NSI) is a Department of Defense measure for symptom presentation and resolution. Reliability and validity are well established. Participants rate 22 symptoms from 0 (not present) to 4 (severe interference with activity). Outcomes include total score and any symptom >1 (yes/no).Total score ranges from 0-88. Assessed at: Initial visit (Baseline); 2 weeks after intervention initiation, determination of asymptomatic state (up to approximately 226 days after intervention initiation); clearance to full return to duty after intervention completion (up to approximately 346 days after intervention initiation).
Quality of Life Perception (PROMIS) | up to approximately 346 days after intervention initiation
  The short version of the PROMIS general scale will be utilized. Participants rate items on scale from 1-5, item scores are summed, and a scale score is computed (range 4-20). Physical function: 4 items (1- unable to do to 5-without any difficulty); anxiety: 4 items (1-never to 5-always); depression: 4 items (1- never to 5-always; fatigue: 4 items (1-not at all to 5-very much); sleep: 4 time (1 to 5); ability to participate in social roles/activities: 4 items (1-always to 5-never); pain interference: 4 items (1-not at all to 5-very much); pain intensity: 1 item (0-no pain to 10-worst pain imaginable). Raw scores are converted to a standardized t-score. Assessed at: Initial visit (Baseline); 2 weeks after intervention initiation, determination of asymptomatic state (up to approximately 226 days after intervention initiation); clearance to full return to duty after intervention completion (up to approximately 346 days after intervention initiation).
Health-related fatigue using the Neuro-QOL Fatigue Scale | up to approximately 346 days after intervention initiation
  Health-related qualify of life fatigue will be assessed using the Quality of Life (QOL) in Neurological Disorders (Neuro-QOL) Fatigue Scale. This scale has reliability and validity concerning overall quality of life. Answers to all 8 items are summed (range 8-40) for a raw summary score. Raw scores are converted to a standardized t-score. Assessed at: Initial visit (Baseline); 2 weeks after intervention initiation, determination of asymptomatic state (up to approximately 226 days after intervention initiation); clearance to full return to duty after intervention completion (up to approximately 346 days after intervention initiation).
Health-related cognition using the Neuro-QOL Cognition Scale | up to approximately 346 days after intervention initiation
  Health-related qualify of life cognition will be assessed using the Quality of Life (QOL) in Neurological Disorders (Neuro-QOL) Cognition Scale. This scale has reliability and validity concerning overall quality of life. Answers to all 8 items are summed (range 8-40) for a raw summary score. Raw scores are converted to a standardized t-score. Assessed at: Initial visit (Baseline); 2 weeks after intervention initiation, determination of asymptomatic state (up to approximately 226 days after intervention initiation); clearance to full return to duty after intervention completion (up to approximately 346 days after intervention initiation).

CONTACTS AND LOCATIONS:
Overall Officials: Johna K Register-Mihalik, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (2):
- United States (2):
  - United States Special Operations Command, Fort Liberty, North Carolina
  - Womack Army Medical Center, Fort Liberty, North Carolina

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared, where allowed by the Department of Defense, beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: IRB, IEC, or REB approval and an executed data use/sharing agreement with UNC, as allowed by the Department of Defense.